CLINICAL TRIAL: NCT00502112
Title: A Phase I Combination Trial of SGN-33 (Anti-huCD33 mAb; HuM195; Lintuzumab) and Lenalidomide (Revlimid®) in Patients With Myelodysplastic Syndromes (MDS)
Brief Title: A Phase I Study of Lintuzumab Combined With Lenalidomide in Patients With Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG033-0002
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Lintuzumab; Antigens, CD33; Antibodies, Monoclonal; Combined Modality Therapy; Myelodysplastic Syndromes; Hematologic Diseases; Preleukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Hematologic Diseases; Preleukemia | interventions — lintuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): lintuzumab and lenalidomide
  Interventions: Drug: lintuzumab; Drug: lenalidomide

INTERVENTIONS:
Drug: lintuzumab — 4 or 8 mg/kg IV (in the vein) on Days 1, 8 and 15 for the first 21-day cycle; 4 or 8 mg/kg IV (in the vein) on Days 1 and 8 for the second through the eighth 21-day cycle
  Other Names: SGN-33
Drug: lenalidomide — 10 or 15 mg per day, taken orally on Days 1-14 of each 21-day cycle
  Other Names: Revlimid

SUMMARY:
This study is a phase I, open-label, single-arm, dose escalation trial to determine the safety and activity of lenalidomide combined with lintuzumab in patients with MDS. Small groups of 3-6 patients will be treated with pre-specified doses of lenalidomide and lintuzumab and will receive 3-week cycles of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Disease confirmation of MDS.
2. Between 5% and 30% blasts in the bone marrow.
3. Received treatment for cytopenias within 2-months
4. ECOG ≤ 2.

Exclusion Criteria:

1. Received prior therapy with lenalidomide, gemtuzumab ozogamicin (Mylotarg®).
2. Received chemotherapy/radiotherapy within 4 weeks of study registration.
3. Received prior bone marrow transplant.
4. 5q- chromosomal deletion in malignant cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events and lab abnormalities | 1 month after last dose

SECONDARY OUTCOMES:
Antitumor activity | Every other 21-day cycle
Pharmacokinetic (PK) profile and immunogenicity (Human Anti-Human Antibody; HAHA) | 1 month after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sievers, MD, Study Director — Seagen Inc.
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - St.Vincent's Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota